CLINICAL TRIAL: NCT03631953
Title: Combination of Alpelisib and Trametinib in Progressive Refractory Meningiomas: Phase 1 Study
Brief Title: Combination of Alpelisib and Trametinib in Progressive Refractory Meningiomas
Acronym: ALTREM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-05; RCAPHM18_0015 (Other: Sponsor's ID)
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — trametinib; Alpelisib; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpelisib in combination with Trametinib administered (Experimental): A panel of 3 doses of Alpelisib could be tested in combination with fixed dose of Trametinib (1.5 mg every day).
  Interventions: Drug: Trametinib; Drug: Alpelisib; Biological: Blood sample; Device: MRI

INTERVENTIONS:
Drug: Trametinib — Trametinib administered at a fixed dose (1.5 mg daily)
Drug: Alpelisib — A panel of 3 doses of ALPELISIB could be tested
Biological: Blood sample — Therapeutic biomarkers
Device: MRI — A MRI with contrast will be performed before treatment start. Assessment of tumor growth.

SUMMARY:
Aggressive growing meningiomas resistant to multiple surgeries and radiotherapy constitute an unmet pharmaceutical need in neurooncology, leading to a fatal issue within a few months. Grade II-III meningiomas progression-free survival (PFS) 6 is at 10-15%. Median PFS grade III meningioma is approximate 3 years.

Alpelisib is a well-tolerated Phosphoinositide 3-kinase α (Pi3Kα) specific inhibitor. However, phosphatidylinositol-3-kinase (PI3K) and the mammalian target of rapamycin (mTOR) inhibition does not induce apoptosis in vitro and induces an antiproliferative effect without any radiologic response in most treated patients.

Trametinib, a mekinist (MEK) inhibitor is currently used in combined treatment for recurrent melanomas in clinical practice with a good clinical tolerance at 1-2 mg daily. In vitro, on meningioma primary cell culture, Trametinib induces cell apoptosis via caspase activity.

These results strongly suggest the relevance to combine Alpelisib and Trametinib in aggressive and recurrent meningiomas.

Alpelisib and Trametinib combination has not been studied to date, despite each drugs have been separately studied in phase 3.

Multicenter, open label, dose-finding phase I study of Alpelisib in combination with Trametinib administered at a fixed dose (1.5 mg daily), both drugs will be administered daily. Starting dose of Alpelisib will be 160mg/day and will be increased to 200mg/day or decreased to 120mg/day depending of grade 3-4 adverse events occurrence, to determine maximal tolerated dose (MTD) and recommended dose.

Primary Objective is to determine the safety profile and tolerability of Alpelisib and Trametinib given in combination in patients with aggressive and refractory meningiomas in terms of Dose-Limiting Toxicities (DLT, assessed during cycle 1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven meningioma grade I, II and III
* Progression is defined as growing meningiomas on 2 different Magnetic Resonance Imaging (MRI) 3 to 6 months apart
* Patients must have failed surgery, and not amenable to a new curative intended surgery
* Patients must have failed radiotherapy and/or radiosurgery
* Patients who have given their written consent
* No contra indication to Alpelisib and Trametinib
* No receiving other investigational agents
* Written informed consent
* Adequate bone marrow function
* Adequate liver function as shown by
* Adequate renal function

Exclusion Criteria:

* Contra indication to Alpelisib and Trametinib
* Women of child-bearing age who are using no effective means of contraception
* Pregnant or breast-feeding women
* Patients receiving other investigational agents
* Known intolerance or hypersensitivity to Alpelisib and Trametinib
* Uncontrolled diabetes mellitus
* Patients who have any severe and uncontrolled medical condition
* Patients receiving chronic treatment with immunosuppressives
* Patients with a known history of HIV seropositivity
* Patients who have a history of another primary malignancy less than or equal to 3 years, with
* the exceptions of non-melanoma skin cancer, and carcinoma in situ of uterine cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) rate of combination Alpelisib and Trametinib | 36 months
  Evaluate adverse events graded (toxicity) according to National Cancer Institute's Common Toxicity Criteria (version 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Oliver ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France